CLINICAL TRIAL: NCT05095155
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: Study of the Prognostic Role of Gene Polymorphism in the Development of B-cell Leukemias and Lymphomas in Children of Kazakh Nationality
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1190
Record Dates: First submitted 2021-10-21; First posted 2021-10-27 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: B Cell Leukemia; Lymphoma
Keywords: SNP
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: children with B-cell leukemia and lymphoma of Kazakhstani nationality
  Interventions: Genetic: SNP analysis of the DNA
- Control group: children without B-cell leukemia and lymphoma of Kazakhstani nationality
  Interventions: Genetic: SNP analysis of the DNA

INTERVENTIONS:
Genetic: SNP analysis of the DNA — SNP analysis of the DNA obtained from peripheral blood sample
  Other Names: SNP analysis of the DNA obtained from peripheral blood sample

SUMMARY:
To search for a genetic marker of B-cell leukemias and lymphomas in children of Kazakh nationality, a single nucleotide polymorphism (SNP) analysis of DNA obtained from the peripheral blood of patients with B-cell leukemias and lymphomas in children of Kazakh nationality and normal control will be performed.

ELIGIBILITY:
Inclusion Criteria:

* ethnicity - Kazakhs in at least three generations
* active disease or a history of B-line ALL or B-NHL, established on the basis of morphological, cytochemical, immunophenotypic or immunohistochemical research methods with confirmation of the fact of the disease in medical documentation
* Signed voluntary informed consent of the legal representative to participate in the project

Exclusion Criteria:

* Children suffering from other types of malignant neoplasms
* Children with B-linear leukemia and lymphomas with concomitant specified genetic and chromosomal diseases
* Children of non-Kazakh nationality
* Absence of signed informed consent or informed refusal of the legal representative to participate in the study before starting therapy

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children of the Kazakh population
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Associated with B-cell lymphoma and B-cell acute lymphoblastic leukemia | 1 year
  Genotype frequency of SNP in the study genes of participants and control participants.

CONTACTS AND LOCATIONS:
Overall Officials: Riza Boranbayeva, PhD, Principal Investigator — JSC "Scientific Center of Pediatrics and Pediatric Surgery"
Locations (1):
- Scientific Center of Pediatrics and Pediatric Surgery, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided